CLINICAL TRIAL: NCT02959723
Title: Physiopathology of Pulmonary Arterial Hypertension: Mechanistic Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Rozenn Quarck, PhD, Clinical Data Manager, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: UZL-S57114; S57114 (Other: UZ Leuven)
Record Dates: First submitted 2015-04-23; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; BMPR2; Inflammation
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Lung tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The current aims to combine analysis of different inflammatory biomarkers and BMPR2 mutations, which are currently analyzed in each patient diagnosed with idiopathic or familial PAH, to establish an earlier diagnosis and consequently better orientate the therapeutic strategy in PAH.

DETAILED DESCRIPTION:
BACKGROUND

Pulmonary hypertension is a severe disorder defined by an elevated mean pulmonary arterial pressure (mPAP) as >25 mmHg at rest. A classification of the different types of pulmonary hypertension has been established according to shared pathologic and clinical features as well as similar therapeutic options and recently updated. Five major categories have been defined including 1) pulmonary arterial hypertension (PAH), 2) PH owing to left heart diseases, 3) PH owing to lung diseases and/or hypoxia, 4) chronic thromboembolic PH (CTEPH) and 5) PH with unclear multifactorial mechanisms.

PAH commonly defined by an elevated PAP (>25 mmHg at rest) and a normal pulmonary arterial wedge pressure (<15 mmHg), is characterized by a pre-capillary arteriopathy with the presence of vascular remodeling and formation of plexiform lesions, an increased pulmonary vascular resistance (PVR), which may result in right heart failure. PAH may be idiopathic (IPAH), heritable (HPAH) or associated with drug/toxin exposure or other medical conditions including connective tissue diseases, congenital heart diseases, human immunodeficiency virus or portal hypertension. Familial cases were already reported in the early fifties and, in 2000, bone morphogenic protein receptor type 2 gene (BMPR2) was identified as the gene responsible for more than 70% of HPAH and about 20% of IPAH. BMPR2 belongs to a superfamily of growth factor receptors, including bone morphogenic protein (BMPs) and transforming growth factor beta (TGF-β) and consequently controls cellular functions such as proliferation, migration, differentiation or apoptosis. BMPR2 mutations may favor activation of p38MAPK-dependent pro-proliferative pathways, which is also ; a key player in cytokine-induced inflammatory signaling pathways. Although BMPR2 mutation carriers develop PAH 10 years earlier than non-carriers and display more severe hemodynamic changes, only 20% of BMPR2 mutation carriers will further develop PAH. A role of inflammation in the pathogenesis of PAH has been suggested. A predictive role of various cytokines has been recently evidenced in PAH. The investigators have observed elevated C-reactive protein (CRP) circulating levels in PAH and evidenced a predictive role of CRP in PAH. Interestingly, heterozygous null BMPR2 mice failed to develop PAH unless an additional inflammatory insult was applied. More recently, inhibition of leukocyte recruitment has been shown to impair PAH progression in mice with genetic ablation of endothelial BMPR-II. This consequently suggests that inflammation could play the role of a second hit in BMPR2 mutation carriers to further develop PAH.

Besides, lipoprotein-associated phospholipase A2 (Lp-PLA2) also named plasma platelet-activating factor-acetylhydrolase (PAF-AH), is the product of PLA2G7 gene and is an enzyme capable of inactivating platelet-activating factor (PAF), a potent lipid mediator of inflammation and a potent vasoconstrictor, and its analogs. Several studies have evidenced an increase in PAF-AH mass and activity in hypercholesterolemia and coronary heart disease. In a recent meta-analysis including more than 70,000 patients from 32 epidemiologic studies, high circulating PAF-AH levels have been identified as an independent predictive risk factor for cardiovascular events. When over-expressed in rodents, Lp-PLA2 displayed anti-inflammatory properties and reduced atherogenesis, suggesting a potential anti-inflammatory role of Lp-PLA2. Lp-PLA2 polymorphisms have been identified and Lp-PLA2 activity has been strongly associated with genetic variants related to LDL- cholesterol levels. In a preliminary study, the investigators have observed a diminished Lp-PLA2 activity in the plasma of PAH patients, together with low total and LDL-cholesterol levels.

HYPOTHESIS & OBJECTIVES

Regarding previous and current results by the investigators, they hypothesized that combining analysis of different inflammatory biomarkers and BMPR2 mutations, which are currently analyzed in each patient diagnosed with idiopathic or familial PAH, could contribute to establish an earlier diagnosis and consequently better orientate the therapeutic strategy. Moreover, BMPR2 gene mutations are responsible for more than 70% of HPAH and about 20% of IPAH; among human BMPR2 mutation carriers, only 20% will further develop PAH, suggesting that BMPR2 mutation itself is not the unique cause for developing PAH and that a second hit, such as inflammation, would be required and play a triggering role in the development of PAH.

METHODOLOGY

1. Identification of biomarkers

   For the current study, one aim is to identify one or several biomarkers which could predict adverse outcome in PAH. To address this aim, the investigators would like to evaluate the levels of CRP, total cholesterol, HDL-cholesterol, triglycerides, albumin, Lp-PLA2 activity, Thrombin Activatable Fibrinolysis Inhibitor (TAFI) and vitamin D in blood plasma from all patients diagnosed with PAH at the UZ Leuven (Campus Gasthuisberg).

   To perform these analyses, the investigators would need 5 tubes of blood:
   * one on EDTA to be sent to the Hospital Laboratory (CRP, lipid profile and albumin);
   * one on citrate to further measure TAFI (Laboratory of Pharmaceutical Biology, KU Leuven);
   * one on EDTA to prepare plasma to be further stored in the laboratory of Pneumology (KU Leuven), from which an aliquot will be sent to INSERM UMRS937 (Paris, France), to measure Lp-PLA2 activity;
   * one on EDTA is sent to the CME genomic DNA isolation to study BMPR2, ALK-1 and ENG mutations; genomic DNA will be stored for potential future genetic;
   * one with Silica Clot Activator to be sent to the Hospital Laboratory (vitamin D).
2. Human pulmonary arterial cell isolation

   Another aim is to investigate whether a relationship between impaired BMPR2 signaling and inflammation could result in dysfunction of pulmonary arterial cells in PAH. To achieve our objective, the investigators propose to investigate:

   i. the in vitro effects of inflammatory mediators and macrophages on the activation of human pre-capillary pulmonary arterial endothelial cell (PAEC) and on the proliferating and migrating properties of PASMC from BMPR2 carriers and non-carriers PAH patients;

   ii. expression and distribution of inflammatory mediators, their receptors and BMPR2 in human lung parenchyma and distal pulmonary arteries;

   iii. the ex-vivo vasoreactive effects of inflammatory mediators mentioned above on isolated human pre-capillary pulmonary arteries.

   iv. Moreover, pulmonary arterial endothelial cells will be harvested from patients undergoing right heart catheterization using a recently described technique, consisting in isolating endothelial cells from the balloon of a Swan-Ganz catheter commonly used to performed right heart catheterization in patients.
3. Pulmonary tissue collection

Lung parenchyma will be collected from i) PAH patients at the time of lung transplantation, ii) eventually unused donor lungs and iii) tissue surrounding lung tumour resection from patients without COPD. Pulmonary pre-capillary endothelial and smooth muscle cells will be isolated, maintained in culture and further stored at low passage number in liquid nitrogen.

Two pieces of lung parenchyma will be snap frozen for further RNA isolation and protein extraction; one piece will be fixed in paraformaldehyde and further processed for immunohistochemistry analyses.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Pulmonary Arterial Hypertension

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Idiopathic Pulmonary Arterial Hypertension undergoing right heart catheterization and/or lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Circulating Inflammatory Biomarkers: CRP, total cholesterol, HDL-cholesterol, triglycerides, albumin, Lp-PLA2 activity, Thrombin Activatable Fibrinolysis Inhibitor (TAFI), vitamin D | Changes from baseline in circulating inflammatory biomarkers will be evaluated at 6 months, 12 months and 24 months whenever a right heart catheterization will be performed after starting a treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided